CLINICAL TRIAL: NCT06657196
Title: The Roles of Critical Closing Pressure and Tissue Perfusion Pressure in Risk Stratification for Patients with Sepsis
Brief Title: Pcrit and TPP for Risk Stratification in Patients with Sepsis
Status: Completed | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Fu Xing Hospital, Capital Medical University (Other); West China Hospital (Other); First Hospital of China Medical University (Other); Shanghai Zhongshan Hospital (Other); The First Hospital of Jilin University (Other); China-Japan Friendship Hospital (Other); Beijing Friendship Hospital of Captial Medical University (Beijing) (Unknown); Beijing Chao Yang Hospital (Other); General Hospital of Ningxia Medical University (Other); Xiangya Hospital of Central South University (Other); Beijing Tongren Hospital (Other); Peking University Third Hospital (Other); Xuanwu Hospital, Beijing (Other); Beijing Tiantan Hospital (Other); Guangdong Provincial People's Hospital (Unknown)
Responsible Party: Sponsor
Other Study IDs: K6349
Record Dates: First submitted 2024-10-08; First posted 2024-10-24 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2024-10

CONDITIONS: Sepsis
Keywords: sepsis; critical closing pressure; tissue perfusion pressure; risk stratification
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: No Intervention: Observational Cohort — No intervention.

SUMMARY:
The goal of this observational study is to learn about the roles of critical closing pressure and tissue perfusion pressure in monitoring hemodynamic status, evaluating organ damage, and predicting mortality risk in patients with sepsis. The main question it aims to answer is:

• Whether increases in critical closing pressure or tissue perfusion pressure are associated with a reduced risk of poor prognosis?

Within the 24 hours following the diagnosis of sepsis, patients will be categorized into four groups based on their 24-hour mean critical closing pressure (Pcc) and tissue perfusion pressure (TPP) estimated from the hourly hemodynamic data within 24 hours. Outcomes will then be compared across these different groups.

The study has been approved by the Medical Ethics Committee of Peking Union Medical College Hospital (K24C1937 and K25C0792).

DETAILED DESCRIPTION:
To validate the reliability of mean Pcc estimated in the primary analysis, we prospectively collected hemodynamic data over a 24-h period from adult ICU patients with invasive arterial monitoring. Two methods were employed to estimate the mean Pcc for reliability validation. Based on the results of preliminary experiment, the sample size calculation showed that at least 12 individuals were needed for reliability validation.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years;
* Sepsis was diagnosed according to Sepsis 3.0 criteria;
* ICU stay exceeding 24 hours after enrollment;
* Undergoing continuous monitoring of vital signs.

Exclusion Criteria:

* Significant absence of blood pressure and heart rate data within 24 hours of enrollment;
* Pregnancy or breastfeeding;
* brain death.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult septic patients who were admitted to ICUs and received continuous monitoring of vital signs.
Sampling Method: Non-Probability Sample
Enrollment: 6769 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
ICU mortality | From the date of trial enrollment until the date of discharge from ICU or date of death from any cause, whichever came first, assessed up to 6 months

SECONDARY OUTCOMES:
In-hospital mortality | From the date of trial enrollment until the date of discharge from hospital or date of death from any cause, whichever came first, assessed up to 6 months
Incidence of acute kidney injury within 7 days of enrollment | From enrollment to 7 days post-enrollment or death
Incidence of acute kidney injury within 48 hours of enrollment | From enrollment to 48 hours post-enrollment or death
The maximum vasoactive inotropic score | From enrollment to 24 hours after enrollment or death

CONTACTS AND LOCATIONS:
Overall Officials: Bin Du, Study Chair — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared upon proper requirement.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After publication of the study.
Access Criteria: Upon proper requirement sent to the primary investigator.

REFERENCES:
- [Background] Evans L, Rhodes A, Alhazzani W, Antonelli M, Coopersmith CM, French C, Machado FR, Mcintyre L, Ostermann M, Prescott HC, Schorr C, Simpson S, Wiersinga WJ, Alshamsi F, Angus DC, Arabi Y, Azevedo L, Beale R, Beilman G, Belley-Cote E, Burry L, Cecconi M, Centofanti J, Coz Yataco A, De Waele J, Dellinger RP, Doi K, Du B, Estenssoro E, Ferrer R, Gomersall C, Hodgson C, Hylander Moller M, Iwashyna T, Jacob S, Kleinpell R, Klompas M, Koh Y, Kumar A, Kwizera A, Lobo S, Masur H, McGloughlin S, Mehta S, Mehta Y, Mer M, Nunnally M, Oczkowski S, Osborn T, Papathanassoglou E, Perner A, Puskarich M, Roberts J, Schweickert W, Seckel M, Sevransky J, Sprung CL, Welte T, Zimmerman J, Levy M. Surviving Sepsis Campaign: International Guidelines for Management of Sepsis and Septic Shock 2021. Crit Care Med. 2021 Nov 1;49(11):e1063-e1143. doi: 10.1097/CCM.0000000000005337. No abstract available. PMID 34605781